CLINICAL TRIAL: NCT00828230
Title: Randomised, Double-blind, Placebo-controlled, Multicentre, Comparative Phase II Pilot Study on the Efficacy and Tolerability of an 8-week Rectal Treatment With 2 mg Budesonide or Placebo for the Prevention of Acute Radiation Proctitis
Brief Title: Budesonide Foam Versus Placebo for Prevention of Acute Radiation Proctitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was prematurely stopped due to slow recruitment after 17 of 32 anticipated patients were recruited.
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BUF-17/RAP; EudraCT No.: 2007-002082-13
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Radiation Proctitis
Keywords: budesonide; placebo; acute radiation proctitis; late radiation proctitis; Prevention of acute radiation proctitis; Prevention of late radiation proctitis
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 2mg rectal budesonide per day for 8 weeks
  Interventions: Drug: budesonide
- 2 (Placebo Comparator): One application of placebo foam once daily for 8 weeks
  Interventions: Drug: Placebo foam

INTERVENTIONS:
Drug: budesonide — One application of 2mg budesonide once daily for 8 weeks
  Other Names: Budenofalk rectal foam
  Arms: 1
Drug: Placebo foam — One application of placebo foam once daily for 8 weeks
  Other Names: placebo
  Arms: 2

SUMMARY:
To proof the superiority of an 8-week rectal treatment with once-daily 2 mg budesonide versus placebo for the prevention of acute radiation proctitis, and to evaluate the occurrence of chronic radiation proctitis 1 year after start of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Men aged at least 18 years,
* Patients with ECOG performance status <= 2 or Karnofsky Performance Status Scale >= 70%,
* Estimated life expectancy more than 3 years,
* Diagnosis of prostate carcinoma,
* Indication for local RT in patients with prostatic cancer.

Exclusion Criteria:

* Crohn's disease, indeterminate colitis, ulcerative colitis, microscopic colitis (i.e., collagenous colitis and lymphocytic colitis),
* Severe or symptomatic ischaemic colitis at baseline,
* Grade III internal haemorrhoids at baseline,
* High risk patients needing extended radiation therapy,
* Acute EORTC/RTOG lower GI toxicity score of >=1 at baseline,
* Bacterial, amoebic, fungal, or viral infections of the gut,
* Tuberculosis, hypertension, infection, diabetes mellitus (included familiarly predisposition), active peptic ulcer, osteoporosis, glaucoma, or cataract, if careful medical monitoring is not ensured,
* Portal hypertension or liver cirrhosis,
* Abnormal hepatic function (ALT, AST or AP > 2.5 x ULN),
* Known intolerance/hypersensitivity/resistance to study drug or drugs of similar chemical structure or pharmacological profile, or to any of the other constituents of the study drug,
* Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients developing radiation proctitis during treatment or need rescue medication | within 8 weeks

SECONDARY OUTCOMES:
Time to occurrence of acute radiation proctitis | During 8 weeks
Time to occurrence of chronic radiation proctitis | Within 1 year
Adverse Events (AEs) | During 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mueller, Dr, Study Director — Dr. Falk Pharma GmbH
Locations (3):
- Germany (3):
  - Klinik für Radioonkologie und Strahlentherapie - Klinikum Braunschweig, Braunschweig
  - Strahlentherapie, St. Vincentius-Kliniken gAG, Karlsruhe
  - Strahlentherapie, Klinikum Mutterhaus der Borromäerinnen, Trier